CLINICAL TRIAL: NCT05728814
Title: A Retrospective, Real-world Multicenter Study of DOstarlimab in Patients With Recurrent or Advanced DNA Mismatch Repair Deficient/Microsatellite Instability-high (dMMR/MSI-H) Endometrial Cancer (DORA Study)
Brief Title: DOstarlimab in Patients With Recurrent or dMMR/MSI-H Endometrial Cancer
Acronym: DORA
Status: Recruiting | Type: Observational
Sponsor: Grupo Español de Investigación en Cáncer de Ovario (Other)
Responsible Party: Sponsor
Other Study IDs: GEICO 120-R & GEICO 120-T
Record Dates: First submitted 2022-12-21; First posted 2023-02-15 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — dostarlimab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Case-only: The study population consists of adult female patients with diagnosis of dMMR/MSI-H recurrent or advanced endometrial cancer with progression to a previous platinum regimen, who were treated within the Spanish dostarlimab Expanded Access Program (EAP).
  Interventions: Drug: Dostarlimab

INTERVENTIONS:
Drug: Dostarlimab — The treatment under observation is dostarlimab administered on day 1 of each treatment cycle until disease progression, unacceptable toxicity or patient/doctor's decision.
  The recommended dose for dostarlimab is 4 cycles of 500 mg every 3 weeks followed by 1000 mg every 6 weeks for all subsequent cycles.

SUMMARY:
This is a multicenter, retrospective, observational (non-interventional) study, in patients treated in a real-world setting within the Spanish dostarlimab EAP. The study is planned to be conducted in the Medical Oncology departments at 50-60 Spanish GEICO-associated hospitals. Its multicenter nature aims to improve the representativeness of the study population in Spain. The study would include approximately 110 patients with dMMR/MSI-H recurrent or advanced EC, that have progressed on or following prior treatment with a platinum containing regimen, treated within the dostarlimab EAP, available in Spain from January 2021 to September 2022. The total number of participating centers and patients will be confirmed once the EAP is closed.

Patient's medical records will be screened by local clinical staff to assess for eligibility according to selection criteria. The study comprises a single study visit, in which the patient will give her informed consent to participate (when the patient is alive) and the physician will extract the study data from the patient's medical charts.

Alive patients who fulfill inclusion criteria and meet no exclusion criteria will be informed by a member of their care team about the purpose of the study, as well as about potential risks and benefits of study participation. The written informed consent form (ICF) should be signed prior to study initiation in alive patients in order to access their medical records. Deceased patients will be still included but their relatives will not be contacted. In these instances, data will be collected by members of the direct care team, unless there is a prior express order from the patient to preserve confidentiality. All eligible deceased and consenting living patients at the participating centers will be included. Data will be directly retrieved from hospital medical records and reported in the electronic Case Report Form (eCRF).

DETAILED DESCRIPTION:
1.1.1. Primary Clinical Objective

• To assess the antitumor activity of dostarlimab in patients with recurrent or advanced mismatch repair deficient (dMMR)/microsatellite instability-high (MSI-H) endometrial cancer, in terms of objective response rate (ORR) and duration of response (DOR) based on investigators' assessment using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

1.1.2. Secondary Clinical Objectives

* To assess the effectiveness of dostarlimab in terms of investigator-assessed progression-free survival (PFS) and overall survival (OS).
* To analyze the PFS rate at 6, 12, 18 and 24 months.
* To assess the disease control rate (DCR) based on investigators' assessment using RECIST 1.1.
* To evaluate duration of treatment with dostarlimab.
* To describe the time to response to dostarlimab.
* To evaluate the safety and tolerability of dostarlimab in patients with dMMR/MSI-H endometrial advanced cancer, including immune-related adverse events of interest (irAEI).
* To evaluate Neutrophil-to-lymphocyte ratio as a potential predictive biomarker for treatment with dostarlimab.

1.1.3. Translational Objectives

* To compare centralized immunohistochemistry (IHC) re-testing with local testing.
* To compare centralized IHC re-testing results with two PCR-based techniques (Promega® and Idylla®) and with possible MMR gene alterations (genetic and epigenetic).
* To analyze the overall response rate and progression-free survival of the dMMR/MSI population selected by each biomarker technique: IHC, Polymerase chain reaction (PCR) Promega®, PCR Idylla®, or gene alteration (next generation sequencing (NGS)/hypermethylation).

1.1.4. Population The study population consists of adult female patients with diagnosis of dMMR/MSI-H recurrent or advanced endometrial cancer with progression to a previous platinum regimen, who were treated within the Spanish dostarlimab Expanded Access Program (EAP)

1.1.5. Treatment Under Observation In this study, the treatment under observation is dostarlimab administered on day 1 of each treatment cycle until disease progression, unacceptable toxicity or patient/doctor's decision.

The recommended dose for dostarlimab is 4 cycles of 500 mg every 3 weeks followed by 1000 mg every 6 weeks for all subsequent cycles.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age, able to understand the program procedures and agree to participate by providing written informed consent.
2. Histologically diagnosed endometrial cancer (note: all histologies are permitted except endometrial sarcoma [including carcinosarcoma]).
3. Patient has evidence of tumor DNA damage repair dysfunction (dMMR/MSI-H) via locally available, validated methodology.
4. Patient has progressed on or after platinum containing chemotherapy (and has received no more than 2 lines of anti-cancer therapy for recurrent or advanced (Stage ≥ IIIB) disease (first or second line)); prior treatment with hormone therapies is acceptable and does not count towards the number of lines of therapy.
5. ECOG performance status of ≤ 2.
6. Adequate organ and bone marrow function, as defined below:

   1. Absolute neutrophil count (ANC) ≥ 1,500/µL
   2. Platelets ≥ 100,000/µL
   3. Hemoglobin ≥ 9 g/dL
   4. Adequate liver and renal function:

      * Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or calculated creatinine clearance ≥ 50 mL/min using Cockcroft-Gault equation for patients with creatinine levels > 1.5 × institutional ULN.
      * Total bilirubin ≤ 1.5 × ULN AND direct bilirubin ≤ 1 × ULN.
      * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN unless liver metastases are present, in which case they must be ≤ 5 × ULN.
7. Cannot be satisfactorily treated with available alternative treatments.
8. Not eligible for a clinical trial with dostarlimab within the indication of the EAP (where access to the clinical trialsite is possible)
9. A female participant is eligible to participate if she is not pregnant or breastfeeding, and if one of the following conditions applies:

   * Is a woman of non-childbearing potential (WONCBP) OR
   * Is a WOCBP and using a contraceptive method that is highly effective (with a failurerate of < 1 % per year), preferably with low user dependency, during treatment and for at least 4 months after treatment. The treating physician should evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated)in relationship to the first doseof dostarlimab.

A WOCBP must have a negative highly sensitive serum pregnancy test within 72 hours before the first dose of dostarlimab. The treating physician is responsible for review of medical history, menstrual history, andrecent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy

Exclusion Criteria:

1. Has received prior therapy with an anti-programmed death-1 (anti-PD-1), anti-PD-1- ligand-1 (anti-PD-L1), or anti-PD-1 ligand-2 (anti-PD-L2) agent.
2. Is considered a poor medical risk due to a serious, uncontrolled medical disorder, non malignant systemic disease, or active infection requiring antibiotic, antifungal or antiviral treatment.
3. Has undergone major surgery 3 weeks prior to initiating dostarlimab (and not recovered from surgical effects).
4. Has malignancies other than endometrial cancer (except for any other malignancy for which the patient is not being actively treated).
5. Has a history of interstitial lung disease.
6. Has an active autoimmune disease that required systemic treatment in the past 2 years (i.e., use of disease-modifying agents, corticosteroids, or immunosuppressive drugs); hormone replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
7. Has experienced ≥ Grade 3 immune related AE with prior immunotherapy, except for non-clinically significant laboratory abnormalities.
8. Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [qualitative] is detected).
9. Has received a live vaccine within 14 days of 1st dose of dostarlimab.
10. Has a known hypersensitivity to dostarlimab components or excipients

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult female patients with diagnosis of dMMR/MSI-H recurrent or advanced endometrial cancer with recurrent disease to a previous platinum, treated within the Spanish dostarlimab EAP.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-04-12 (Estimated); Study Completion 2024-09-12 (Estimated)

PRIMARY OUTCOMES:
Dostarlimab Treatment | Month 4-6
  End of treatment reason (toxicity, doctor's decision, patient's decision, progression or other)
Dostarlimab Treatment | Month 4-6
  Number of cycles Number of interruptions
Dostarlimab Treatment | Month 4-6
  Start date (first dose) End of treatment date
Disease progression after dostarlimab | Month 4-6
Best Response Assessment | Month 4-6
Dostarlimab -Related Adverse Events | Month 4-6

SECONDARY OUTCOMES:
Demographics | Month 4-6
Medical History | Month 4-6
Endometrial Cancer History | Month 4-6
Endometrial Cancer Previous Treatments | Month 4-6
Baseline (pre-dostarlimab) | Month 4-6
Death | Month 4-6
Survival Status | Month 4-6
Subsequent Therapies for Endometrial Cancer | Month 4-6

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Gallego Martinez, Principal Investigator — Clinica Universitaria de Navarra; Marta Mendiola Sabio, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Arnau de Vilanova, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT05728814/Prot_000.pdf